CLINICAL TRIAL: NCT01704300
Title: Body Mass Index and Initial Presentations of Cardiovascular Diseases
Acronym: CALIBER
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Principal Investigator, Harry Hemingway, Harry Hemingway, FRCP, University College, London
Other Study IDs: CALIBER 10_14
Record Dates: First submitted 2012-10-08; First posted 2012-10-11 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Abdominal Aortic Aneurysm; Acute Myocardial Infarction; Stroke; Heart Failure; Peripheral Arterial Disease; Angina
Keywords: Abdominal aortic aneurysm; Acute Myocardial Infarction; Coronary heart disease not otherwise specified; Haemorrhagic stroke; Heart failure; Ischaemic stroke; Peripheral arterial disease; Stable angina; Unheralded coronary death; Unstable angina; Ventricular arrhythmias, cardiac arrest and sudden cardiac death; Transient Ischemic Attack
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Stroke; Heart Failure; Peripheral Arterial Disease; Angina Pectoris; Hemorrhagic Stroke; Ischemic Stroke; Angina, Stable; Angina, Unstable; Heart Arrest; Death, Sudden, Cardiac; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CALIBER Healthy Cohort: We will report findings from the CALIBER (CArdiovascular disease research using Linked BEspoke studies and Electronic Records) collaboration where we linked primary care data (from the General Practice Research Database [GPRD]) to three further sources of electronic health records: the Myocardial Ischemia National Audit Project registry (MINAP),cause specific discharge data from Hospital Episodes Statistics (HES) and cause specific mortality from the Office for National Statistics (ONS).

SUMMARY:
The association between obesity and cardiovascular disease (CVD) has mostly been studied using broad endpoints or have focused on cause-specific mortality. The investigators aim to compare the effect of body mass index (BMI) on different types of initial presentation of CVD.

DETAILED DESCRIPTION:
Obesity has many detrimental effects on the cardiovascular system that can manifest in a range of clinical presentations. Many of these are mediated by frequently coexisting conditions such as diabetes, hypertension and dyslipidemia but there are also direct, progressive effects on the arteries and the heart muscle. As evident from autopsies, even from early adulthood the degree of coronary artery disease (CAD) correlates with the BMI and particularly the amount of abdominal fat. The multiple mechanisms by which obesity exerts its effects are still being elucidated.

Previous studies have assessed the effect of obesity on cause-specific mortality. Here the investigators analyze association of BMI with the first symptomatic presentation of cardiovascular disease across any phenotypes, to which the investigators refer to as "initial presentation" to distinguish from first presentation within a specific phenotype. For example, an initial presentation with myocardial infarction is an MI which is not preceded by stable angina, ischemic stroke or any other phenotype, rather than the first MI in a possible series of MIs, as is commonly used in other studies.

Adjustments The key risk factor of interest is baseline BMI, which the investigators define as the most recent measurement of BMI recorded up to 2 years prior to cohort entry date. BMI will be analyzed based on the following categories: underweight (<18.5 kg/m2), healthy (18.5 to 24 kg/m2), overweight (25 to 29 kg/m2), moderately obese (30 to 34 kg/m2), morbidly obese (>35 kg/m2). The healthy BMI category will be used as the reference in regression models.

Associations with BMI will be adjusted for age, sex, ethnicity, social deprivation, smoking, diabetes, and systolic blood pressure, total cholesterol (TCHOL) and high-density lipoprotein cholesterol (HDL). All baseline covariates will be obtained from within a 2 year window prior to study entry.

Statistical analyses Cause-specific Cox models will be used to measure the association between BMI categories and endpoints of interest. Multiple imputation will be used to replace missing values in prognostic factors. The investigators will estimate lifetime risk for each endpoint over time adjusting for competing risks.

ELIGIBILITY:
Inclusion Criteria:

* Baseline age ≥30 years

Exclusion Criteria:

* prior atherosclerotic disease or stroke

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The cohort we will use in the present analysis has been drawn from patients across 225 practices in England contributing data to GPRD, covering approximately 5% of the UK population (Figure 1). The study period is 1st January 2001 to 25th March 2010 (the date of the last GPRD data submission). To allow time for medical history and risk factors to be measured and recorded we require that patients enter the cohort after having completed at least 1 year of registration with their current practice during which the practice provides data that meet research quality criteria. Patients are followed up from the date they become eligible to be included in the cohort until the earliest date among a) the date of an initial presentation with one of the endpoints of interest, b) the date of leaving the practice or c) the date of last data submission from their practice.
Sampling Method: Non-Probability Sample
Enrollment: 2240000 (Actual)
Dates: Start 2001-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University College London, London, United Kingdom